CLINICAL TRIAL: NCT02343289
Title: An Open-Label Study to Evaluate the Absolute Bioavailability of Intranasal and Oral Esketamine and the Effects of Clarithromycin on the Pharmacokinetics of Intranasal Esketamine in Healthy Subjects
Brief Title: A Study to Evaluate the Absolute Bioavailability of Intranasal and Oral Esketamine and the Effects of Clarithromycin on the Pharmacokinetics of Intranasal Esketamine in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR106240; ESKETINTRD1009 (Other: Janssen Research & Development, LLC); 2014-004055-31 (EudraCT Number)
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Healthy; Pharmacokinetics; Esketamine; JNJ-54135419
MeSH Terms: interventions — Esketamine; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Esketamine Regimen (Experimental): All participants will first receive 28 milligram (mg) of esketamine as a single, 40-minute, intravenous infusion on Day 1 of Period 1, followed by 84 mg of esketamine solution as a single, oral dose on Day 1 of Period 2, followed by 84 mg of intranasal esketamine on Day 1 of Period 3 and then 500 mg of clarithromycin twice daily on Days -3, -2, -1, 1, and 2 of Period 4 and 84 mg of intranasal esketamine on Day 1 of Period 4. Each period will be separated by a washout period of up to 21 days in between.
  Interventions: Drug: Esketamine; Drug: Clarithromycin

INTERVENTIONS:
Drug: Esketamine — 28 mg of esketamine as a single, 40-minute, intravenous infusion on Day 1 of Period 1, 84 mg of esketamine solution as a single, oral dose on Day 1 of Period 2, 84 mg of intranasal esketamine on Day 1 of Period 3 and on Day 1 of Period 4.
Drug: Clarithromycin — 500 mg of clarithromycin twice daily on Days -3, -2, -1, 1, and 2 of Period 4.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of esketamine administered by the intranasal (administered through the nose) and oral routes and to evaluate the effects of clarithromycin on the pharmacokinetics of intranasally administered esketamine.

DETAILED DESCRIPTION:
This is a single-center, 4-period, fixed-sequence, open-label study. The study consists of Screening Period (Days -21 to -2), Open-label Treatment Period 1, 2, 3, 4 and End of Study (9 to 13 days after final dose or at Early Withdrawal). The total duration of study will be up to 98 days. For all 4 periods, the participants will be admitted into the study center on Day -1 of each treatment period and receive a 28 milligram (mg) (intravenous) or 84 mg (oral and intranasal) esketamine dose regimen on Day 1 of each period in a fixed sequence. Participants will also receive 500 mg of clarithromycin in period 4. Blood samples will be collected to evaluate the pharmacokinetic parameters. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* For women of childbearing potential, must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at screening; and a negative urine pregnancy test on Day -1 of Period 1
* If a man, must agree to use an adequate contraception method as deemed appropriate by the investigator (example, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Participants with body mass index (BMI) between 18 and 30 kilogram per square meter (kg/m^2) (inclusive), and body weight not less than 50 kg
* Participants with blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic
* Participants should be comfortable with self-administration of intranasal medication and able to follow instructions provided

Exclusion Criteria:

* Participants diagnosed with a psychiatric disorder including but not limited to psychotic, bipolar, major depressive, or anxiety disorder
* Participants with clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic disease, infection, hypertension or vascular disorders, kidney or urinary tract disturbances, sleep apnea, myasthenia gravis, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participants with clinically significant abnormal values for hematology, clinical chemistry (particularly potassium or magnesium levels below the normal laboratory range), or urinalysis at screening or at admission to the study center (Day -1 of Period 1) as deemed appropriate by the investigator
* Participants with clinically significant abnormal physical examination and vital signs at screening or at admission to the study center (Day -1 of Period 1) as deemed appropriate by the investigator
* Participants with history of drug or alcohol abuse disorder within the past 1 year, or a reason to believe a participant has such a history

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Esketamine | Pre-dose, 0.25, 0.33, 0.5, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48 hr post-dose on Day 3 in all periods
  The Cmax is the maximum plasma concentration.
Time to Reach Maximum Plasma Concentration (Tmax) of Esketamine | Pre-dose, 0.25, 0.33, 0.5, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48 hr post-dose on Day 3 in all periods
  The Tmax is time to reach the maximum plasma concentration.
Area Under the Plasma Concentration-time Curve From Time 0 to 12 Hours (AUC12h) of Esketamine | Pre-dose, 0.25, 0.33, 0.5, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hour (hr) post-dose on Day 1 in all periods
  The (AUC12h) is the area under the plasma concentration-time curve from time 0 to 12 hours Post-dose.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time of the Last Quantifiable Concentration AUC(0-last) of Esketamine | Pre-dose, 0.25, 0.33, 0.5, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48 hr post-dose on Day 3 in all periods
  The (AUC [0-last]) is the area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of Esketamine | Pre-dose, 0.25, 0.33, 0.5, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48 hr post-dose on Day 3 in all periods
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(0-last)/lambda(z), wherein AUC(0-last) is the area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentrations; C(0-last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Percentage of Area Under the Plasma Concentration-time Curve Obtained by Extrapolation (%AUC [infinity,ex]) of Esketamine | Pre-dose, 0.25, 0.33, 0.5, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48 hr post-dose on Day 3 in all periods
  Percentage of area under the plasma concentration-time curve obtained by extrapolation (%AUC[inf,ex]) is calculated by dividing the difference of AUC(0-infinity) and AUC(0-last) by AUC(0-infinity) and then multiplying by 100 (AUC[0-infinity] - AUC[0-last])*100/AUC[0-infinity].
Elimination Half-life (t1/2) of Esketamine | Pre-dose, 0.25, 0.33, 0.5, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48 hr post-dose on Day 3 in all periods
  Elimination half-life (t [1/2]) is associated with the terminal slope (lambda [z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Rate Constant (Lambda[z]) of Esketamine | Pre-dose, 0.25, 0.33, 0.5, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48 hr post-dose on Day 3 in all periods
  Lambda(z) is first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Absolute Bioavailability (Fabs) of Esketamine | Pre-dose, 0.25, 0.33, 0.5, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48 hr post-dose on Day 3 in all periods
  The absolute bioavailability (Fabs) based on AUC(0-last) and AUC(0-inf) and estimated as 100*Test/Reference, where Test is defined as the pharmacokinetic parameters of oral esketamine and intranasal esketamine without clarithromycin and Reference is defined as intravenous esketamine.
Relative Bioavailability of Esketamine (Frel) | Pre-dose, 0.25, 0.33, 0.5, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 hour (hr) post-dose on Day 1; 24, 36 hr post-dose on Day 2; 48 hr post-dose on Day 3 in all periods
  The relative bioavailability (Frel) based on Cmax, AUC(0-last), and AUC(0-inf) and estimated as 100*Test/Reference, where Test is defined as the pharmacokinetic parameters of intranasal esketamine and Reference is defined as intranasal esketamine + clarithromycin.
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | Throughout the duration of study (approximately up to 98 days)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium

REFERENCES:
- [Derived] Perez-Ruixo C, Rossenu S, Zannikos P, Nandy P, Singh J, Drevets WC, Perez-Ruixo JJ. Population Pharmacokinetics of Esketamine Nasal Spray and its Metabolite Noresketamine in Healthy Subjects and Patients with Treatment-Resistant Depression. Clin Pharmacokinet. 2021 Apr;60(4):501-516. doi: 10.1007/s40262-020-00953-4. Epub 2020 Oct 31. PMID 33128208